CLINICAL TRIAL: NCT02218255
Title: Eeva™ Pregnancy Pilot Study (PPS)
Acronym: PPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Progyny, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013-AUX-010
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Infertility
Keywords: In Vitro Fertilization
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Day 3 eSET combined with Eeva (Active Comparator): Traditional Morphology + Eeva™ results
  Interventions: Device: Eeva™ results
- Day 5 eSET combined with Eeva (Active Comparator): Traditional Morphology + Eeva™ results
  Interventions: Device: Eeva™ results
- Day 5 eSET with Traditonal Morphology (No Intervention)

INTERVENTIONS:
Device: Eeva™ results
  Arms: Day 3 eSET combined with Eeva; Day 5 eSET combined with Eeva

SUMMARY:
The purpose of this clinical investigation is to gather pilot data to evaluate the impact of using Eeva™, a time-lapse enabled embryo test, in combination with traditional morphology on clinical pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing fresh in vitro fertilization treatment using their own eggs
* ≤ 40 years
* ≥ 4 diploid embryos (i.e. having 2 PNs)
* ≤ 3 Prior ART cycles (IVF, ICSI and related procedures)
* All 2PN embryos (for all 3 arms) must be imaged by Eeva
* Subject willing to comply with study protocol and procedures
* Subject willing to provide written informed consent

Exclusion Criteria:

* Preimplantation genetic diagnosis or preimplantation genetic screening
* Planned "freeze all" cycle (eggs or embryos)
* Asherman's Syndrome
* Donor egg
* Gestational carrier
* Presence of Hydrosalpinx on ultrasound
* Concurrent participation in an interventional clinical study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy | 7-8 weeks gestation

SECONDARY OUTCOMES:
Ongoing pregnancy rate | 8-12 week gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kaser DJ, Bormann CL, Missmer SA, Farland LV, Ginsburg ES, Racowsky C. A pilot randomized controlled trial of Day 3 single embryo transfer with adjunctive time-lapse selection versus Day 5 single embryo transfer with or without adjunctive time-lapse selection. Hum Reprod. 2017 Aug 1;32(8):1598-1603. doi: 10.1093/humrep/dex231. PMID 28854588